CLINICAL TRIAL: NCT02907437
Title: Minocycline add-on Medication to Antipsychotics in the Treatment of Schizophrenia Patients: A Double- Blind Randomized Controlled Trial
Brief Title: Minocycline add-on to Antipsychotics for the Treatment of Negative and Cognitive Symptoms in Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beer Yaakov - Ness Ziona Mental Health Center (Other Government)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Dr. Stryjer Rafael (MD), Senior Psychatrist, Beer Yaakov - Ness Ziona Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 519
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: Minocycline; Negative symptoms; Cognitive symptoms; Inflammation
MeSH Terms: conditions — Schizophrenia; cyclopia sequence; Neurobehavioral Manifestations; Inflammation | interventions — Minocycline; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minocycline treatment (Active Comparator): Intervention: Drug: Minocycline (200 mg/day)
  Interventions: Drug: Minocycline; Other: Probiotics
- Placebo treatment (Placebo Comparator): Placebo Intervention: Drug: Placebo (200 mg/day)
  Interventions: Drug: Placebo; Other: Probiotics

INTERVENTIONS:
Drug: Minocycline — Minocycline as an add-on drug (200 mg/day)
  Arms: Minocycline treatment
Drug: Placebo — (200 mg/day)
  Arms: Placebo treatment
Other: Probiotics — (450 mg/day)

SUMMARY:
Current medications have only a limited effect on two core symptoms of schizophrenia, negative symptoms and cognitive deficits. Minocycline is a second-generation tetracycline which has a beneficial effect in various neurological disorders. In the past years, various findings from clinical studies showed its potential role for the treatment of these symptoms of schizophrenia. The current study aims to examine the efficacy of minocycline as add-on treatment for alleviating positive, negative and cognitive symptoms in schizophrenia patients.The current study is a single center, double-blind, randomized study that assess the adjuvant therapeutic effect of minocycline vs. placebo added to antipsychotic medications, in adult patients suffering from schizophrenia. Patients will be recruited and randomly allocated to a minocycline or placebo treatment (200 mg/day) for 6 weeks of treatment. In addition, all patients will receive probiotics (450mg/day) in order to prevent any gastrointestinal influences of antibiotics administration. Positive and negative symptoms , as well as cognitive functions will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-60 years of age.
2. Diagnostic and Statistical Manual (DSM) 5 diagnosis of Schizophrenia/ Schizo effective disorder based on the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID) for schizophrenia and confirmed by two senior psychiatrists.
3. Initiated on treatment with stable dosage (within +/- 25%) of atypical anti-psychotic medication for at least 6 weeks.
4. Capable and willing to provide informed consent.
5. Able to adhere to the treatment schedule.
6. Able to read, hear, write and speak the local language.
7. Has signed a written informed consent to participate in the study.

Exclusion Criteria:

1. Patients with acute, unstable, or decompensated medical condition.
2. Present substance abuse.
3. Major depression (MDD) diagnosis.
4. Attention deficit/ hyperactivity disorder (ADHD/ADD) diagnosis.
5. Cognitive dysfunction, such as Alzheimer disease or retardation.
6. Acute psychotic state.
7. Aggressive or violent patient or with vast history of aggressive or violent behavior.
8. Diagnosis of Borderline/ Anti Social/ Narcissistic personality disorders.
9. Previous sensitivity to Minocycline.
10. Current suicidal ideation or history of a suicide attempt in the past three years
11. Known or suspected pregnancy or women of childbearing potential not using a medically accepted form of contraception .(if using oral contraceptives, during the Minocycline treatment, subject should use an additional contraceptives), or women who are breastfeeding.
12. Subjects who are taking a known contraindication to Minocycline treatment (anti-coagulants, other antibiotics (of the penicillin group), methoxyflurane, Isotretinoin).
13. Subjects who had received treatment with Minocycline or β-lactam antibiotics in the preceding half year before study entry.
14. Subjects who are under compulsory hospitalization.
15. Subjects with medical history of Intestinal disease, Peptic ulcer or gastritis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-02 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Change in PANSS scores over the 6-weeks study
Scale for Assessment of Negative Symptoms (SANS) | Change in SANS scores over the 6-weeks study

SECONDARY OUTCOMES:
Clinical Global Impressions (CGI) | Change in CGI scores over the 6-weeks study
The Montreal Cognitive Assessment (MoCa) task | Change in MoCa scores over the 6-weeks study
Trail making task (TMT) | Change in TMT scores over the 6-weeks study
Empathy Cartoon task | Change in Empathy Cartoon task scores over the 6-weeks study
Interpersonal Reactivity Index (IRI) Questionnaire | Change in IRI scores over the 6-weeks study

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Stryjer, MD, Principal Investigator — Beer Yaakov - Ness Ziona Mental Health Center
Locations (1):
- Bees Yaakov and Ness Ziona Mental Health Center, Beer Yaakov, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chaudhry IB, Hallak J, Husain N, Minhas F, Stirling J, Richardson P, Dursun S, Dunn G, Deakin B. Minocycline benefits negative symptoms in early schizophrenia: a randomised double-blind placebo-controlled clinical trial in patients on standard treatment. J Psychopharmacol. 2012 Sep;26(9):1185-93. doi: 10.1177/0269881112444941. Epub 2012 Apr 23. PMID 22526685
- [Background] Chaves C, de Marque CR, Wichert-Ana L, Maia-de-Oliveira JP, Itikawa EN, Crippa JA, Zuardi AW, Todd KG, Baker GB, Dursun SM, Hallak JE. Functional neuroimaging of minocycline's effect in a patient with schizophrenia. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Apr 16;34(3):550-2. doi: 10.1016/j.pnpbp.2010.01.020. Epub 2010 Feb 6. No abstract available. PMID 20138948
- [Background] Davis MC, Horan WP, Marder SR. Psychopharmacology of the negative symptoms: current status and prospects for progress. Eur Neuropsychopharmacol. 2014 May;24(5):788-99. doi: 10.1016/j.euroneuro.2013.10.010. Epub 2013 Nov 4. PMID 24252823
- [Background] Dean OM, Data-Franco J, Giorlando F, Berk M. Minocycline: therapeutic potential in psychiatry. CNS Drugs. 2012 May 1;26(5):391-401. doi: 10.2165/11632000-000000000-00000. PMID 22486246
- [Background] Jhamnani K, Shivakumar V, Kalmady S, Rao NP, Venkatasubramanian G. Successful use of add-on minocycline for treatment of persistent negative symptoms in schizophrenia. J Neuropsychiatry Clin Neurosci. 2013 Winter;25(1):E06-7. doi: 10.1176/appi.neuropsych.11120376. No abstract available. PMID 23487204
- [Background] Khodaie-Ardakani MR, Mirshafiee O, Farokhnia M, Tajdini M, Hosseini SM, Modabbernia A, Rezaei F, Salehi B, Yekehtaz H, Ashrafi M, Tabrizi M, Akhondzadeh S. Minocycline add-on to risperidone for treatment of negative symptoms in patients with stable schizophrenia: randomized double-blind placebo-controlled study. Psychiatry Res. 2014 Mar 30;215(3):540-6. doi: 10.1016/j.psychres.2013.12.051. Epub 2014 Jan 9. PMID 24480077
- [Background] Levkovitz Y, Mendlovich S, Riwkes S, Braw Y, Levkovitch-Verbin H, Gal G, Fennig S, Treves I, Kron S. A double-blind, randomized study of minocycline for the treatment of negative and cognitive symptoms in early-phase schizophrenia. J Clin Psychiatry. 2010 Feb;71(2):138-49. doi: 10.4088/JCP.08m04666yel. Epub 2009 Nov 3. PMID 19895780
- [Background] Monji A, Kato T, Kanba S. Cytokines and schizophrenia: Microglia hypothesis of schizophrenia. Psychiatry Clin Neurosci. 2009 Jun;63(3):257-65. doi: 10.1111/j.1440-1819.2009.01945.x. PMID 19579286
- [Background] Lisiecka DM, Suckling J, Barnes TR, Chaudhry IB, Dazzan P, Husain N, Jones PB, Joyce EM, Lawrie SM, Upthegrove R, Deakin B. The benefit of minocycline on negative symptoms in early-phase psychosis in addition to standard care - extent and mechanism (BeneMin): study protocol for a randomised controlled trial. Trials. 2015 Mar 2;16:71. doi: 10.1186/s13063-015-0580-x. PMID 25886254
- [Background] Meyer U, Schwarz MJ, Muller N. Inflammatory processes in schizophrenia: a promising neuroimmunological target for the treatment of negative/cognitive symptoms and beyond. Pharmacol Ther. 2011 Oct;132(1):96-110. doi: 10.1016/j.pharmthera.2011.06.003. Epub 2011 Jun 15. PMID 21704074